CLINICAL TRIAL: NCT02338622
Title: A Phase I Multi-centre Trial of the Combination of Olaparib (PARP Inhibitor) and AZD5363 (AKT Inhibitor) in Patients with Advanced Solid Tumours
Brief Title: Trial of Olaparib in Combination with AZD5363 (ComPAKT)
Acronym: ComPAKT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4058; 2013-004692-13 (EudraCT Number)
Record Dates: First submitted 2014-07-03; First posted 2015-01-14 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2020-01

CONDITIONS: Advanced Cancer
Keywords: olaparib; AZD5363; intrapatient dose escalation; advanced solid tumours
MeSH Terms: interventions — olaparib; capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schedule A: 4 days on, 3 days off (Experimental): 300mg olaparib + intrapatient dose escalation of AZD5363 4 days on, 3 days off
  Schema for dose escalation in schedule A (4-days-on, 3-days-off AZD5363)
  -1. Olaparib: 200mg, AZD5363 240mg
  1. Olaparib: 300mg, AZD5363 320mg
  2. Olaparib: 300mg, AZD5363 400mg
  3. Olaparib: 300mg, AZD5363 480mg
  Interventions: Drug: olaparib; Drug: AZD5363
- Schedule B: 2 days on, 5 days off (Experimental): 300mg olaparib + intrapatient dose escalation of AZD5363 2 days on, 5 days off
  Schema for dose escalation in schedule B (2-days-on, 5-days-off AZD5363)
  -1. Olaparib: 200mg, AZD5363 400mg
  1. Olaparib: 300mg, AZD5363 480mg
  2. Olaparib: 300mg, AZD5363 560mg
  3. Olaparib: 300mg, AZD5363 640mg
  Interventions: Drug: olaparib; Drug: AZD5363

INTERVENTIONS:
Drug: olaparib — olaparib BD
  Other Names: AZD2281
Drug: AZD5363 — AZD5363 BD

SUMMARY:
This is a phase I trial of the combination of the PARP inhibitor olaparib and AKT inhibitor AZD5363.

There are two parts to this study. Part A: dose escalation, and Part B: dose expansion.

Part A will investigate the combination of 300 mg bd of olaparib with intrapatient ascending doses of AZD5363 administered for either 4-days-on, 3-days-off, and 2-days-on, 5-days-off.

Once the Maximum Tolerated Dose (MTD) is reached for both arms (or under the advice from the Safety Review Committee (SRC) one of the schedules will be discontinued), the schedule with the optimum safety and PK/PD profile will be taken forward to a dose expansion phase (Part B).

Part B will evaluate the optimized dose/schedule identified in Part A of the study in patients with (1) BRCA1/2 mutant cancers (with previous disease progression on PARP inhibitor monotherapy), or (2) advanced sporadic tumours (e.g. TNBC, CRPC, HGSOC and tumours with somatic mutations or other aberrations known to result in a hyperactivated PI3K-AKT pathway).

DETAILED DESCRIPTION:
Part A: The starting doses for both intermittent schedules will be 300 mg bd of olaparib and either AZD5363 given at 320 mg bd 4-days-on, 3-days-off, or 480 mg bd 2-days-on, 5-days-off. These starting doses are based on available data from the first-in-human studies [D0810C00002] (AstraZeneca) and [D3610C00001] (AstraZeneca) of both drugs, respectively.

A general schema for 3 potential dose levels to be pursued on the 4-days-on, 3-days-off AZD5363 schedule (Schedule A) and 2-days-on, 5-days-off AZD5363 schedule (Schedule B) in Part A of the study are listed below. The starting dose of olaparib will be fixed at 300mg bd in both schedules. These schema only provide general guidance; it will be possible for doses of one or both drugs to be escalated or de-escalated in a "seesaw" fashion contingent on the toxicity and/or PK/PD data reported. This may create dose cohort combinations not listed below. Both PK and PD data will be taken into consideration if available. With the exception of dose level 1, actual dose escalation/de-escalation will be determined following a discussion with the SRC during dose escalation teleconferences. Dose escalation will continue until MTD(s) are reached. Patients will be dosed on a flat scale and not by body weight or body surface area. Both schedules will be carried out in parallel.

Table 1: Schema for dose escalation in schedule A (4-days-on, 3-days-off AZD5363) Dose level (DL) olaparib bd AZD5363 bd 4d-on, 3d-off

* 1 200mg* 240mg

  1. 300mg 320mg
  2. 300mg 400mg
  3. 300mg 480mg

     *An intermediate dose of 250mg bd of olaparib may be considered depending on drug-related toxicities observed and patient tolerability

     Table 2: Schema for dose escalation in schedule B (2-days-on, 5-days-off AZD5363) Dose level (DL) olaparib bd AZD5363 bd 2d-on, 5d-off
* 1 200mg* 400mg

  1. 300mg 480mg
  2. 300mg 560mg
  3. 300mg 640mg

     * An intermediate dose of 250mg bd of olaparib may be considered depending on drug-related toxicities observed and patient tolerability

After careful review of the clinical toxicity data, if the DLT is deemed to be caused by one of the agents, the responsible drug may be dose decreased and if well tolerated, the other agent maybe be increased in subsequent cohorts. If necessary, both drugs can also be dose de-escalated.

In Part A of the study, olaparib will be administered continuously with intermittent AZD5363 in 21-day cycles. Intrapatient dose escalation of AZD5363 will be utilised to evaluate different dose levels. The optimal dose schedule selected based on toxicity, PK-PD and/or efficacy data will be taken forward into two expansion cohorts in Part B of the study. Cohort 1 will comprise patients with germline BRCA1/2 mutated tumours, while Cohort 2 will comprise advanced sporadic cancers that may harbour HR defects (e.g. TNBC, CRPC and HGSOC) or those with somatic mutations or other aberrations known to result in a hyperactivated phosphatidylinositol-3-kinase (PI3K)-AKT pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Part A: Patients with histologically or cytologically confirmed malignant advanced solid tumours refractory to standard therapy or for which no suitable effective standard therapy exists, including, but not limited to patients with: BRCA1/2 mutant cancers, TNBC, CRPC and HGSOC, and those with somatic mutations or other aberrations known to result in a hyperactivated PI3K-AKT pathway.

   Part B: (1) BRCA1/2 mutation cohort: Patients with advanced germline BRCA1/2 mutant solid tumours; (2) Sporadic cancers cohort: This cohort will include advanced sporadic cancers that are not known to harbour germline BRCA1/2 mutations, but which may harbour homologous recombination (HR) defects, e.g. advanced TNBC, CRPC and HGSOC, and those with somatic mutations or other aberrations known to result in a hyperactivated PI3K-AKT pathway.
2. Life expectancy of at least 12 weeks
3. WHO performance status of 0-1 with no significant deterioration over the previous 2 weeks
4. Evaluable or measurable disease as assessed by RECIST 1.1
5. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week.

   * Hb ≥ 10.0 g/dL
   * Absolute neutrophil count ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Serum bilirubin ≤ 1.5 x upper limit of normal except for patient with documented Gilburt's disease
   * ALT or AST ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 times ULN is permissible

If creatinine > 1.5 times ULN then: Either:

* Creatinine Clearance ≥ 50 mL/min (uncorrected value)
* Isotope clearance measurement ≥ 50 mL/min (corrected) 6.18 years or over 7. Signed and dated informed consent and be capable of co-operating with treatment and follow-up

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) and 4 weeks for investigational medicinal products before treatment, except for hormonal therapy with luteinizing hormone-releasing hormone analogues for medical castration in patients with CRPC, which are permitted.
2. Ongoing toxic manifestations of previous treatments. Exceptions to this are Grade 1 toxicities, which in the opinion of the Investigator should not exclude the patient.
3. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.
4. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
5. Major surgery (excluding minor procedures, e.g. placement of vascular access) within 4 weeks of the first dose of study treatment.
6. At high medical risk because of severe or uncontrolled systemic disease including active bleeding diathesis or active infection including hepatitis B, hepatitis C and human immunodeficiency virus. Screening for chronic conditions is not required.
7. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

   * Diagnosis of diabetes mellitus type I or II (irrespective of management).
   * HbA1C ≥ 8.0% at screening (64 mmol/mol) (conversion equation for HbA1C [IFCC-HbA1C (mmol/mol)] = [DCCT-HbA1C (%) - 2.15] x 10.929)
   * Fasting Plasma Glucose ≥ 8.9mmol/L at screening. Fasting is defined as no caloric intake for at least 8 hours.
8. Proteinuria 3+ on dipstick analysis or >500mg/24 hours.
9. Previous treatment with a PARP inhibitor or PI3K/AKT inhibitor (Part B: sporadic cancers arm of dose expansion cohort only).
10. Treatment with potent inhibitors or inducers or substrates of CYP3A4 or substrates of CYP2D6 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort).
11. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment
12. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 consecutive electrocardiograms
    * Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
    * Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association [NYHA0 Grade 2
    * Uncontrolled hypotension - Systolic BP <90mmHg and/or diastolic BP <50mmHg
    * LVEF below institutional lower limit of normal.
13. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of olaparib and AZD5363.
14. History of hypersensitivity to active or inactive excipients of AZD5363 or olaparib or drugs with a similar chemical structure or class to AZD5363 and olaparib.
15. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study. Participation in an observational trial would be acceptable.
16. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
17. Patients with myelodysplastic syndrome or acute myeloid leukaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability of olaparib in combination with AZD5363 | 3 to 9 weeks at least.
  Dose at which no more than one out of six patient at the same dose level experiences a probable drug-related dose limiting toxicity.
Maximum tolerated dose and recommended Phase II dose of this combination in patients with advanced solid tumours. | 3 to 9 weeks at least.
  Dose at which no more than one out of six patient at the same dose level experiences a probable drug-related dose limiting toxicity.

SECONDARY OUTCOMES:
Plasma levels of olaparib and AZD5363 using validated assays. | Average of 2 years
  Plasma levels of olaparib and AZD5363 using validated assays.
pAkt/Akt, pGSK/GSK3, pS6 kinase/S6 kinase and pPRAS40/PRAS40 ratios in pre- and post-treatment tumour biopsies using validated assays. | Average of 2 years
  Changes in platelet rich plasma, hair follicles and pre- and post-treatment tumour biopsies using validated assays

OTHER OUTCOMES:
Exploratory biomarkers | Average of 2 years
  Changes in exploratory biomarkers, including pERK, RAD51, BRCA and PARP expression in pre- and post-treatment tumour biopsies
Putative predictive biomarkers of response and resistance in archival tumours and fresh tumour biopsies | Average of 2 years
  Correlate anti-tumour activity of the combination of olaparib and AZD5363 with the detection of putative predictive biomarkers of response and resistance in archival tumours and fresh tumour biopsies
Disease response by RECIST criteria v1.1 and tumour markers and change in tumour size | Average of 2 years
  Preliminary assessment of the antitumour putative predictive biomarkers of response and resistance to the combination of olaparib and AZD5363.
MTD safely established using an intrapatient dose escalation strategy | Average of 2 years
  Evaluate a novel experimental trial design involving intrapatient dose escalation of AZD5363 in combination with olaparib.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Yap, MBBS MRCP PhD, Principal Investigator — The Institute of Cancer Research, The Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Northern Institute for Cancer, Freeman Hospital, Newcastle, Newcastle upon Tyne
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey

REFERENCES:
- [Background] Yap TA, Kristeleit R, Michalarea V, Pettitt SJ, Lim JSJ, Carreira S, Roda D, Miller R, Riisnaes R, Miranda S, Figueiredo I, Rodrigues DN, Ward S, Matthews R, Parmar M, Turner A, Tunariu N, Chopra N, Gevensleben H, Turner NC, Ruddle R, Raynaud FI, Decordova S, Swales KE, Finneran L, Hall E, Rugman P, Lindemann JPO, Foxley A, Lord CJ, Banerji U, Plummer R, Basu B, Lopez JS, Drew Y, de Bono JS. Phase I Trial of the PARP Inhibitor Olaparib and AKT Inhibitor Capivasertib in Patients with BRCA1/2- and Non-BRCA1/2-Mutant Cancers. Cancer Discov. 2020 Oct;10(10):1528-1543. doi: 10.1158/2159-8290.CD-20-0163. Epub 2020 Jun 12. PMID 32532747